CLINICAL TRIAL: NCT00251264
Title: Arthroscopic Versus Open Stabilization of Traumatic Unidirectional Anterior Shoulder Instability: A Randomized Clinical Trial
Brief Title: Arthroscopic Versus Open Stabilization for Traumatic Shoulder Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Calgary Regional Health Authority (CRHA) (Other Government); Calgary Orthopaedic Research and Education Fund (Other); Canadian Orthopaedic Foundation (Other)
Responsible Party: Principal Investigator, Dr. Nicholas Mohtadi, Clinical Professor and Orthopaedic Surgeon, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15740
Record Dates: First submitted 2005-11-08; First posted 2005-11-09 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Joint Instability; Shoulder Dislocation
Keywords: Shoulder instability; Traumatic; Anterior; Unidirectional; Open stabilization; Arthroscopic; Bankart repair; Shoulder instability, traumatic; Anterior, unidirectional instability; Bankart
MeSH Terms: conditions — Joint Instability; Shoulder Dislocation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open (Active Comparator)
  Interventions: Procedure: Open stabilization
- Arthroscopic (Active Comparator)
  Interventions: Procedure: Arthroscopic stabilization

INTERVENTIONS:
Procedure: Open stabilization — Following examination under anesthesia, a 5cm standard deltopectoral incision is made. Dissection is continued exploiting the deltopectoral internervous plane. The conjoined tendon is retracted medially. The underlying subscapularis tendon is identified and incised horizontally or split vertically in its midsubstance. If required for adequate exposure, the subscapularis split may be extended by incising the inferior component of the subscapularis tendon near its insertion on the lesser tuberosity. The shoulder is entered by performing a "T" shaped arthrotomy with retractors for full exposure of the glenoid. Shoulder pathology is addressed with suture anchor repair of any capsulolabral detachment (ie.Bankart lesion) and/ or a capsular plication for repair of capsular redundancy.
  Other Names: open shoulder stabilization; open Bankart reconstruction
  Arms: Open
Procedure: Arthroscopic stabilization — With the examination under anesthesia completed, the arthroscope is introduced through a standard posterior arthroscopy portal. A diagnostic arthroscopy is performed and the intraarticular pathology identified and documented. Any labral detachment (i.e. Bankart lesion) is repaired using suture anchor fixation and arthroscopic tying techniques. Capsular redundancy is addressed with the use of thermal electrocapsulorrhaphy or arthroscopic suture repair of the redundant capsule. With the repair complete, 40 cc of 0.5% Bupivicaine is introduced into the joint. A sterile dressing is applied over the wounds and the operated shoulder placed in a shoulder immobilizer.
  Other Names: Scope stabilization; Arthroscopic reconstruction
  Arms: Arthroscopic

SUMMARY:
The purpose of this study is to compare arthroscopic and open shoulder stabilization procedures by measuring the disease-specific quality of life outcome in patients with traumatic unidirectional anterior instability of the shoulder at 2 and 5 years.

Hypothesis: There is no difference in disease-specific quality of life outcomes in patients with traumatic unidirectional anterior shoulder instability, undergoing an arthroscopic versus an open stabilization procedure.

DETAILED DESCRIPTION:
Shoulder instability most commonly affects people in the late teens to mid thirties, which are the most active years, recreational and vocational. The resulting disability, time lost from work, as well as the effect on an individual's quality of life represent a significant clinical problem for the population and for the healthcare system.

The normal anatomy in the unstable shoulder can be restored using arthroscopic or open surgical stabilization techniques. There is considerable controversy surrounding the issue of arthroscopic versus open shoulder stabilization. Advocates of arthroscopic procedures cite the following as advantages: faster recovery, less post operative pain, decreased operative time, improved cosmetics, greater return of shoulder motion and the more accurate identification of intraarticular pathology. Those in favor of an open procedure cite superior long term results showing fewer recurrences with an open stabilization.

There are few published reports directly comparing arthroscopic versus open shoulder stabilization repairs. It is also difficult to compare the results of existing studies as they report on heterogeneous patient populations, using a variety of techniques on mixed pathologies, using different outcome scales and variable definitions of success and failure. This study will address this controversial issue by comparing the disease-specific quality of life outcomes in patients with traumatic unidirectional anterior shoulder instability undergoing an arthroscopic versus an open stabilization procedure.

This study is designed as a prospective randomized clinical trial with a second prospective analytical cohort study arm. In the randomized arm, patients are assigned to arthroscopic or open surgery based on varied block, computer-generated randomization. The expertise-based randomization method is used in this study, whereby the surgeons perform either arthroscopic or open surgery, but not both. Therefore, a patient is not only randomized to a treatment group, but is also assigned to the expert surgeon for that treatment.

Patients in the prospective analytical cohort study arm of the trial undergo shoulder stabilization (open or arthroscopic) with any surgeon and complete the same follow-up visits, however they have not been randomized. The outcomes of the prospective cohort will be compared to those of the randomized arm to determine if the expertise-based randomization method has an effect on patient outcome.

Disease-specific quality of life is assessed using the validated Western Ontario Shoulder Instability (WOSI) Index. The index has 21 questions divided into 4 categories: physical symptoms, sport/recreation/work, lifestyle and emotions. This self-administered questionnaire utilizes a 100mm visual analog scale format to provide an overall score out of 100. A lower score reflects a better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Clinical:

  * Age 14 years or greater
  * Diagnosis of traumatic anterior shoulder instability, made by meeting all of the following:

    1. Radiographic evidence or documented physician assisted reduction of anterior shoulder dislocation following a traumatic injury.
    2. Ability to elicit unwanted glenohumeral translation which reproduce symptoms with one of the following tests: anterior apprehension, relocation test, or anterior load and shift test
* Radiological:

  * Closed growth plate on a standardized series of x-rays consisting of a minimum of an anteroposterior view, lateral in the scapular plane and an axillary view.

Exclusion Criteria:

* Clinical:

  * Diagnosis of multidirectional instability (MDI) or multidirectional laxity with anteroinferior instability (MDL-AII), made by two or more of:

    1. Symptomatic (pain or discomfort) in inferior or posterior direction
    2. Ability to elicit unwanted posterior glenohumeral translation that reproduces symptoms with posterior apprehension tests, or posterior load and shift test
    3. Positive sulcus sign of 1cm or greater that reproduces patient's clinical symptoms
  * Previous surgery on the affected shoulder other than diagnostic arthroscopy
  * Cases involving litigation
  * Significant tenderness of acromioclavicular/sternoclavicular joints on affected side
  * Confirmed connective tissue disorder (ie: Ehlers-Danlos, Marfan)

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2001-11; Primary Completion 2010-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Western Ontario Shoulder Instability (WOSI) Index | Baseline, 3, 6, 12, 24 months post-operatively

SECONDARY OUTCOMES:
American Shoulder and Elbow Society (ASES) score | Baseline, 3, 6, 12, 24 months post-operatively
Physical examination: range of motion, strength, stability | Baseline, 3, 6, 12, 24 months post-operatively
Return to sport or activity, return to work | Baseline, 3, 6, 12, 24 months post-operatively
Complications | Intra-operatively and up to 2 weeks post-operatively
Time to perform each procedure | Day of surgery
Economic cost of each procedure | Day of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Mohtadi, MD, FRCSC, Principal Investigator — University of Calgary Sport Medicine Centre; Robert Hollinshead, MD, FRCSC, Principal Investigator — University of Calgary Sport Medicine Centre
Locations (1):
- University of Calgary Sport Medicine Centre, Calgary, Alberta, Canada

REFERENCES:
- [Background] Kirkley A, Griffin S, Richards C, Miniaci A, Mohtadi N. Prospective randomized clinical trial comparing the effectiveness of immediate arthroscopic stabilization versus immobilization and rehabilitation in first traumatic anterior dislocations of the shoulder. Arthroscopy. 1999 Jul-Aug;15(5):507-14. doi: 10.1053/ar.1999.v15.015050. PMID 10424554
- [Background] McLAUGHLIN HL, CAVALLARO WU. Primary anterior dislocation of the shoulder. Am J Surg. 1950 Nov 15;80(6):615-21; passim. doi: 10.1016/0002-9610(50)90581-2. No abstract available. PMID 14790098
- [Background] Rowe CR, Patel D, Southmayd WW. The Bankart procedure: a long-term end-result study. J Bone Joint Surg Am. 1978 Jan;60(1):1-16. PMID 624747
- [Background] Arciero RA, Wheeler JH, Ryan JB, McBride JT. Arthroscopic Bankart repair versus nonoperative treatment for acute, initial anterior shoulder dislocations. Am J Sports Med. 1994 Sep-Oct;22(5):589-94. doi: 10.1177/036354659402200504. PMID 7810780
- [Background] Green MR, Christensen KP. Magnetic resonance imaging of the glenoid labrum in anterior shoulder instability. Am J Sports Med. 1994 Jul-Aug;22(4):493-8. doi: 10.1177/036354659402200410. PMID 7943514
- [Background] Kirkley A, Griffin S, McLintock H, Ng L. The development and evaluation of a disease-specific quality of life measurement tool for shoulder instability. The Western Ontario Shoulder Instability Index (WOSI). Am J Sports Med. 1998 Nov-Dec;26(6):764-72. doi: 10.1177/03635465980260060501. PMID 9850776
- [Background] Hawkins RB. Arthroscopic stapling repair for shoulder instability: a retrospective study of 50 cases. Arthroscopy. 1989;5(2):122-8. doi: 10.1016/0749-8063(89)90007-8. PMID 2736008
- [Background] Morgan CD, Bodenstab AB. Arthroscopic Bankart suture repair: technique and early results. Arthroscopy. 1987;3(2):111-22. doi: 10.1016/s0749-8063(87)80027-0. PMID 3300681
- [Background] Baker CL, Uribe JW, Whitman C. Arthroscopic evaluation of acute initial anterior shoulder dislocations. Am J Sports Med. 1990 Jan-Feb;18(1):25-8. doi: 10.1177/036354659001800104. PMID 2301687
- [Background] Cash JD. Recent advances and perspectives on arthroscopic stabilization of the shoulder. Clin Sports Med. 1991 Oct;10(4):871-86. PMID 1934102
- [Result] Mohtadi NG, Chan DS, Hollinshead RM, Boorman RS, Hiemstra LA, Lo IK, Hannaford HN, Fredine J, Sasyniuk TM, Paolucci EO. A randomized clinical trial comparing open and arthroscopic stabilization for recurrent traumatic anterior shoulder instability: two-year follow-up with disease-specific quality-of-life outcomes. J Bone Joint Surg Am. 2014 Mar 5;96(5):353-60. doi: 10.2106/JBJS.L.01656. PMID 24599195